CLINICAL TRIAL: NCT05215522
Title: Upper Limb Telerehabilitation Using Brain -Controlled Functional Electrical Stimulation
Brief Title: Tele BCI-FES for Upper -Limb Stoke Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sheffield (Other)
Collaborators: Sheffield Teaching Hospitals NHS Foundation Trust (Other); Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: USheffield1
Record Dates: First submitted 2021-12-13; First posted 2022-01-31 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2021-12

CONDITIONS: Stroke
Keywords: Brain-computer interface; functional electrical stimulation; Tele-rehabilitation; stroke rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The BCI-FES Intervention (Experimental): The BCI-FES device will be used by all participants.
  Interventions: Device: The BCI-FES Intervention

INTERVENTIONS:
Device: The BCI-FES Intervention — To evaluate whether the participant can effectively control FES using the developed remote BCI system. Thus, participants will receive a three-week BCI-FES intervention at their home, including three sessions of intervention per week. Each session will last around 60 minutes, including 10 minutes of preparation, 40 minutes of intervention and 10 minutes interview on the user's experience with the device and any experienced side effects, if any.

SUMMARY:
The study aims to identify whether stroke survivors can intentionally modulate their brain signals for controlling an FES device to produce arm movements for home based rehabilitation. The study also assess the participants acceptability of this new home-based rehabilitation.

DETAILED DESCRIPTION:
Movements of different parts of the body, including the arm, start when the brain produces specific electrical signals. Sometimes after a stroke, even though the person intends to move the arm, the arm will not move or will only move partly. The brain continues to produce electrical signals after stroke, but when the signals are weak the arm does not move. Brain-computer interface (BCI), is a method of utilising the brain signals to produce useful outputs via computers. One type of BCI is BCI Functional Electrical Stimulus (BCI-FES) which is a device that can detect these brain signals produced during the intention to move the weak arm after a stroke. It then uses these signals to trigger an electrical stimulator. The electrical stimulator then stimulates the muscles in the weak arm to produce the desired arm movement. Recent studies show that rehabilitation using this device has given better results when compared with conventional rehabilitation approaches. However, the BCI-FES devices currently available are bulky and participants need to come to the hospital or laboratory to receive the treatment. Our project aims to develop a BCI-FES device, called Tele BCI-FES that can be used at stroke participant's home. The investigators are using techniques like machine learning to make the Tele BCI-FES quick and simple to set up, easy to use and effective. This study aims to investigate if the proposed Tele BCI-FES device is a feasible and acceptable intervention for post-stroke rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

1) Age 18 and above.

(2) Experienced an ischaemic or haemorrhagic stroke more than 6 months ago.

(3) Arm weakness interfering with activities of daily living.

(4) Fugl-Meyer score of upper limb<45.

(5) Caregiver is willing to assist with trial by helping to deliver intervention.

(6) Cognitive and language abilities to understand and participate in the study protocol.

(7) Can maintain sitting with or without support for 1 hour continuously.

(8) Able to give consent and understand instructions.

Exclusion criteria:

1. Cognitive impairment that would interfere with their ability to comply with the experimental protocol or provide informed consent;
2. Dermatological, rheumatologic or orthopaedic illnesses of the affected arm interfering with movement of the elbow;
3. Pre-existing severe systemic disorders like cardiovascular disease; active cancer or renal disease; end stage pulmonary or cardiovascular disease; psychiatric illness including severe alcohol or drug abuse
4. Inability to perform the baseline assessments;
5. Severe tactile hypersensitivity;
6. Participation in other, upper limb rehabilitation studies
7. Within 12 weeks of receiving Botulinum toxin injections;
8. History of epilepsy
9. Pace maker or any other implanted devices
10. Pregnancy
11. Severe dystonia/spasm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Evaluate the feasibility of the proposed system through the ability of participants to control the Tele BCI-FES | within 10 minutes after experimental session
  To evaluate whether the participants can effectively control FES using the developed remote BCI system (Success: the BCI accuracy of more than 70% in at least 7 out of 9 sessions).
Evaluate the usability and acceptability of the proposed system based on the number of participants completing each TeleBCI-FES intervention session | through study completion, an average of 5 weeks
  Number of participants completing each TeleBCI-FES intervention session (Success: 7 participants completed 8 or more of 12 TeleBCI-FES sessions)
Recruitment rate | Pre-intervention
  To measure the acceptability of the proposed rehabilitation

SECONDARY OUTCOMES:
Fugl-Meyer Assessment | Pre-intervention and up to 5 weeks
  It is the most frequently used outcome scales to measure post stroke motor recovery of the upper extremity on a scale of 0-60 (best).
Action Research Arm Test | Pre-intervention and up to 5 weeks
  It is a 19 item observational measure used to assess upper extremity performance on a scale of 0 - 57 (best).
Modified Ashworth Scale | Pre-intervention and up to 5 weeks
  This looks at elbow and wrist flexors on predefined scale. The scale ranges from 0 to 4 (worst).
Medical Research Council grading | Pre-intervention and up to 5 weeks
  This looks at assessing muscle strength from Grade 5 (normal) to Grade 0 (no visible contraction) and takes around 10 minutes to complete.
Leeds Arm Spasticity Scale-reference | Baseline and up to 5 weeks
  It is a measure of passive arm function, suitable for participants with spasticity and little or no active movement of the upper extremity. The score ranges from 0 (No difficulty) to 4 (Inability to perform the activity).
Numerical rating Scale (NRS) | Pre-intervention and up to 5 weeks
  It requires the participant to rate their pain on a defined scale from 0 (no pain) to 10 (the worst pain)
Pittsburgh Participation in Rehabilitation scale | within 10 minutes after experimental session
  It is a clinician-rated measure on a 6-point Likert-type scale that quantifies individuals' participation in their therapy sessions, ranging from 1 (None: participant refused the entire session) to 6 (Excellent: participant participated in all sessions)
European Quality of List 5D-5L (EQ-5D-5L): | Pre-intervention and .up to 5 weeks
  It is a self-assessed, health related, quality of life questionnaire. The scale measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each level is assigned a rating based on the severity of the problems in that area (no problems walking, minor problems, moderate problems, severe problems, or inability to walk). The tool also includes an overall health scale, on which the participant chooses a number between 1 and 100 (best) to represent their health status.

OTHER OUTCOMES:
Interviews | within 10 minutes after experimental session
  A qualitative assessment of the effectiveness and acceptability of treatment for participants.

CONTACTS AND LOCATIONS:
Overall Officials: Mahnaz Arvaneh, PhD, Principal Investigator — University of Sheffield
Locations (1):
- Sheffield Teaching Hospitals, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The participant's data will be "pseudo-anonymized" and no identifiable information will be maintained with the study data because the participant will be issued a unique study number. Paper copies of consent forms will be kept in locked cupboards at the University of Sheffield's Physiological Signals and Systems lab. Electronic data will be entered and saved immediately on a password-protected University server. After the study is completed, anonymised EEG data and questionnaire data will be preserved for fifteen years at the University of Sheffield archiving facility. The results of this study will be published in peer-reviewed journals. The findings will be presented in BCI and rehabilitation conferences, as well as patient-public involvement meetings. The participants will not be identifiable from any report or publication placed in the public domain.

REFERENCES:
- [Derived] Mansour S, Giles J, Nair KPS, Marshall R, Ali A, Arvaneh M. A clinical trial evaluating feasibility and acceptability of a brain-computer interface for telerehabilitation in patients with stroke. J Neuroeng Rehabil. 2025 Apr 24;22(1):91. doi: 10.1186/s12984-025-01607-x. PMID 40269846
- See also: A website introducing our technology, and our team — https://teleregain.com/